CLINICAL TRIAL: NCT00374374
Title: Treatment With Lactobacillus Rhamnosus and Lactobacillus Acidophilus for Patients With Active Colonic Crohn's Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19990156
Record Dates: First submitted 2006-09-07; First posted 2006-09-11 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-04

CONDITIONS: Crohn's Disease
Keywords: probiotic
MeSH Terms: conditions — Crohn Disease

INTERVENTIONS:
Behavioral: Administration of probiotic

SUMMARY:
The purpose of this study is to determine whether a probiotic containing Lactobacillus Acidophilus and Lactobacillus Rhamnosus is effective as treatment for patients with active colonic Crohn's disease

DETAILED DESCRIPTION:
The aetiology of Crohn's disease is still not known. In the recent years there has been an increasing interest in the relationship between the gastrointestinal flora and gut function. Several studies have shown promising results for the use of probiotics in patient with inflammatory bowel disease.

Aim: The aim of the current study is to evaluate the effect of a probiotic suspension in patients with active colonic Crohn's disease.

Methods: The study is a two-centre, randomised placebo-controlled, and double-blind trial. Patients above the age of 18 years, attending our out-patient clinic, can be included if they have Crohn's disease in the colon or colon and small bowel and have active disease with a CDAI: 220-400. Patients are not included if they have undergone larger bowel resections, have been treated with antibiotics within the last two months, if dose of prednisolone has been changed within the last 4 weeks, or dose of immunosuppressives has been changed within the last 2 months. During the study period no changes in medication is allowed. During an 8 week period patients are treated with a combination of lactobacillus rhamnosus strain 19070-2 and lactobacillus acidophilus strain 18911-2 (10EE9 colony forming unit/ml). Freeze-dried probiotics are dissolved in sterile water to a volume of 1 ml which is ingested once daily, in the evening.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed Crohn's disease of the large bowel or large and small bowel according to established criteria.
* At least one prior episode of active disease
* Stoolcultures and microscopies without pathogenic bacteria or parasites
* CDAI 220-400
* Informed consent

Exclusion Criteria:

* More than 15mg of prednisolone daily (or equivalent)
* Changes in dosage of glucocorticoids during the last four weeks prior to inclusion
* Changes in dosage of Azathioprine during the last 3 months prior to inclusion
* Antibiotic treatment during the last two months prior to inclusion
* Symptoms of Crohn's disease assumed to be caused by mechanical obstruction og abscesses
* Long term treatment with NSAID or colestyramine
* Pregnant and lactating women
* Bowel resections removing more than 100 centimetres of small intestine or any colonic resection other than ileo-cecal resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2001-05; Study Completion 2005-11

PRIMARY OUTCOMES:
Decrease in CDAI

SECONDARY OUTCOMES:
Increase in IBDQ

CONTACTS AND LOCATIONS:
Overall Officials: Lone G Klinge, Principal Investigator — Odense University Hospital; Jens Kjeldsen, MD, PhD, Principal Investigator — Odense University Hospital; Karsten Lauritsen, Study Chair — Odense University Hospital; Ole Oestergaard-Thomsen, Principal Investigator — Herlev Hospital
Locations (1):
- Dept. of Medical Gastroenterology (afd.S), Odense University Hospital, Odense, Denmark